CLINICAL TRIAL: NCT04953689
Title: Technology-assisted Conscientiousness Therapy for People With Multiple Sclerosis
Acronym: TACT-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Ralph H.B. Benedict, Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003473
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis
Keywords: neuropsychology; multiple sclerosis; conscientiousness; mobile application; smartphone application; employment; quality of life
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: One group is assigned the intervention, one group is assigned to a waitlist control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Conscientiousness Coach
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: Conscientiousness Coach — Participants will use the Conscientiousness Coach app to organize their goals and assist them in engaging in more conscientious behaviors. The participant will also be educated about Conscientiousness as it relates to healthy living and accomplishing life goals and values. Participants will receive brief phone calls during weeks 1, 2, 6, and 10 from the research assistant, tracking progress, answering queries, and return visits to the clinic/teleconference will be scheduled for further assistance during week 4 and week 8. These mid-study visits (or 'Booster Sessions') will last approximately 50 minutes and will involve a brief discussion of goal and value progress and app usage; at this in-person meeting/teleconference, similar questions and topics will be covered as in the bi-monthly phone calls. At week 12, there is a treatment termination visit with the principal investigator and research assistant.
  Other Names: C.Coach; C.App
  Arms: Intervention

SUMMARY:
This is a validation study of a conscientiousness-based phone app intervention strategy to help people with their health management and employment.

DETAILED DESCRIPTION:
The primary objective is to establish whether people with MS with low Conscientiousness benefit from a cognitive-behavioral, phone app intervention. Also enrolled are healthy individuals over the age of 60. This group's response to the intervention will be compared to the MS sample. The investigators also aim to determine the acceptability and utilization of the Conscientiousness-Coach phone application and intervention. It is anticipated that the Conscientiousness-Coach phone app intervention will result in fewer negative work events and increased work accommodations in those treated, relative to the control group. In exploration of other secondary outcomes, the investigators also expect that the treatment will result in increased self-report trait Conscientiousness itself, increase in structured leisure activities, reduction in depression, and reduction in anxiety.

This is a prospective longitudinal design with an experimental manipulation (i.e., a randomized-controlled trial). There will be an initial assessment with neuropsychological testing, the Buffalo Vocational Monitoring Survey (BVMS), and several self-report measures, and a post-test assessment after three months and six months with these same instruments, excluding the neuropsychological assessment. The BVMS will also be administered at 0 months, 3 months, and 6 months to further assess post-treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of Multiple Sclerosis or is over 60 years of age.
* If an MS patient: is above 18 years of age.
* No history of substance dependence/abuse, psychiatric disorders, or any neurological disease other than MS
* If an MS patient: has a NEO-FFI Conscientiousness score that is one standard deviation or more below the healthy adult mean (t=40)

Exclusion Criteria:

• Does not meet one or more of the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Self -Reflection and Insight Scale (SRIS): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24.
  20 question self-report measure which assesses participants private self-consciousness using self-reflection and insight components. Total score of 20-120 points is calculated, with higher scores indicating greater self-reflection and insight.
Buffalo Vocational Monitoring Survey (BVMS): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24
  Assesses general employment information (e.g. number of hours worked per week, job title, and income) and work-related problems and accommodations. Participants will identify specific negative work events (e.g. formal reprimand) experienced in the past 3 months and provide a list of job accommodations to endorse if they are receiving them at the time of survey. Income, number of hours worked per week, number of negative work events (0 to 7, with higher number indicating more negative work events), and number of accommodations (0 to 40, with higher number indicating more accommodations) will be used as outcomes from this survey.
The Valued Living Questionnaire (VLQ): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24
  Assesses valued living, or the extent to which an individual contacts his or her chosen values in everyday life. Respondents are asked to rate the 10 areas of life on a scale of 1-10, indicating the level of importance and how consistently they have lived in accord with those values in the past week. The composite score is used (1-100 points), with higher scores indicating a greater extent to which one is living out particular values in everyday life.

SECONDARY OUTCOMES:
NEO Five Factor Inventory (NEOFFI): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24.
  Personality inventory measuring five primary domains of personality: neuroticism, extraversion, openness, agreeableness, and conscientiousness. Total scores are 12-60 on each domain's scale, with higher scores indicating higher levels of that personality trait.
Quality of Life in Neurological Disorders (NeuroQol): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24.
  Measure of quality of life for neurology patients. We are using the four subscales of Communication, Ability to Participate in Social Roles and Activities, Satisfaction with Social Roles and Activities, and Positive Affect and Well Being. T-scores are used with higher T-scores indicating greater quality of life in each respective domain.
Beck Depression Inventory 2nd Edition (BDI-II): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24.
  Quantifies depression symptoms. Minimum of 0, maximum of 63. Higher score indicates higher levels of depression.
Beck Anxiety Inventory (BAI): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24.
  Quantifies anxiety symptoms. Minimum of 0, maximum of 63. Higher score indicates higher levels of anxiety.
Multiple Sclerosis Work Difficulties Questionnaire (MSWDQ-23): change from baseline to 12 weeks and from baseline to 24 weeks | At baseline, Week 12, and Week 24.
  Measures work-related problems in multiple sclerosis patients. Scale of 0-100 with higher scores indicating greater work difficulty.
The Symbol Digit Modalities Test (SDMT) | At baseline only
  Presents a series of nine symbols, each paired with a single digit in a key at the top of a stimulus page. Subjects voice the number associated with each symbol as rapidly as possible. Measures cognitive processing speed. Minimum score of 0, Maximum score of 120. Higher scores indicate better performance.
The California Verbal Learning Test Second Edition (CVLT2) | At baseline only
  Measures verbal learning and memory. Begins with the examiner reading a list of 16 words. Patients listen to the list and report as many of the items as possible. After recall is recorded, the entire list is read again followed by a second attempt at recall. Altogether, there are five learning trials, and a delayed recall trial after 20 minutes. Minimum of 0, maximum of 80 on learning trials. Minimum of 0, maximum of 16 on delayed recall trial. Higher score indicates better performance.
The Brief Visuospatial Memory Test Revised (BVMTR) | At baseline only
  Measures visual/spatial memory. Presents six abstract designs for 10 seconds. The display is removed from view and patients render the stimuli via pencil on paper manual responses. There are three learning trials and a delayed recall trial after 20 minutes. Minimum of 0, maximum of 36 on learning trials. Minimum of 0, maximum of 12 on delayed recall trial. Higher score indicates better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Conventus Building, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuchs TA, Jaworski MG 3rd, Youngs M, Abdel-Kerim O, Wojcik C, Weinstock-Guttman B, Benedict RHB. Preliminary Support of a Behavioral Intervention for Trait Conscientiousness in Multiple Sclerosis. Int J MS Care. 2022 Mar-Apr;24(2):45-53. doi: 10.7224/1537-2073.2021-005. Epub 2021 Jul 9. PMID 35462870